CLINICAL TRIAL: NCT05969145
Title: The Effect of Hot-Cold Application to the Bladder After Orthopedic Surgery on Postoperative Urinary Retention
Acronym: PUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Elif Demirden Erişti, Principal investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ankara Bilkent Sehir Hastanesi
Record Dates: First submitted 2023-05-10; First posted 2023-08-01 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Urinary Retention
Keywords: orthopedic surgery; hot-cold application; postoperative urinary retention

STUDY DESIGN:
Intervention Model Description: a single-blind randomized controlled trial to determine the effect of hot-cold application to the bladder on postoperative urinary retention in orthopedic surgery patients.
Who Masked: Participant
Masking Description: The participant will not know that there is a control or experimental group. The result evaluator is an independent statistical expert, and the data analysis will be performed by a statistical specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hot-cold application (Experimental): This group will be given a hot cold application to the bladder
  Interventions: Procedure: application of thermophor
- control group (No Intervention): Routine clinical functioning will be applied to this group

INTERVENTIONS:
Procedure: application of thermophor — The experimental group will be given hot and cold application to the bladder
  Arms: hot-cold application

SUMMARY:
The development of postoperative urinary retention (PUR) is a significant complication in patients undergoing treatment due to orthopedic surgery. In particular, it is reported that the incidence rate of PUR after spinal anesthesia is in the range of 6-60%. It is stated in the literature that PUR can be prevented by reviewing factors such as bladder physical examination, fluid intake status, anesthesia type, bladder discharge time/condition of patients undergoing orthopedic surgery. For this purpose, our study showed that these patients had globular physical examination screening and postoperative 2-6. it aims to prevent postoperative urinary retention by applying hot and cold Decontamination to the bladders of patients who cannot urinate spontaneously between hours.

DETAILED DESCRIPTION:
Orthopedic surgery is a surgical treatment method based on the correction of the functions of bones, November muscles, tendons, and ligaments in the body. Arthroplasty (hip, knee, shoulder), arthroscopy (meniscopathy, rotator cuff rupture), limb fractures, structural (hallux vagus, hallux rigidities, carpal tunnel syndrome, trigger finger), and developmental (hip dysplasia) dysfunctions are the interventions in which the orthopedic surgical procedure is performed. In orthopedic surgeries, the need for surgical treatment increases every day as a result of degeneration in the musculoskeletal system with a decrease in mobilization due to advancing age, November illness, trauma, or technological developments. In the United States, 30% of major surgical interventions involve orthopedic surgeries performed on elderly individuals); in Turkey, it is reported that 33.5% of orthopedic surgeries are performed due to trauma, and about 48% are performed on the lower extremities. Orthopedic surgeries are practices that risk serious complications, as with any treatment option. Complications such as nausea, vomiting, headache, hypotension, and postoperative urinary retention (PUR), especially due to spinal anesthesia, may be observed in patients receiving treatment due to orthopedic surgery. While the prevalence of PUR in orthopedic surgeries is 6-40% in the literature, it is stated that this rate is higher (6-60%) after spinal anesthesia. Due to PUR after orthopedic surgery, there is an increase in hospital stay times, susceptibility to infection, deterioration in the quality of life, and associated cost increases.

Postoperative urinary retention is a complication that manifests symptoms with problems such as suprapubic pain, bladder spasm, and/or inability to urinate after surgical treatment. The etiology of PUR includes factors caused by the patient (advanced age, male gender, anatomical problems, comorbidity, neural transmission disorders), due to the surgical process (failure to empty the bladder during the preoperative period, surgery lasts longer than 2 hours, emergency surgery, opioid-NSAID-atropine use, amount of fluid taken) and due to anesthesia (epidural/spinal anesthesia). 2-6 of the postoperative period. it gives symptoms as a result of the absence of the first urine decrement between hours. As a result, serious problems such as increased urinary pressure and acute kidney injury and/or dysfunction due to bladder distension occur in patients. Management of PUR can be achieved by using physical examination (globe monitoring), bladder catheterization, and ultrasonographic (USG) methods to diagnose these problems at an early stage.

Field health professionals, who have an important place in the conduct of health services, offer the greatest contribution to the surgical treatment process with their understanding of quality health care. In particular, nurses who are actively involved in the perioperative process are the professional staff with the greatest responsibility for positively managing health care. Nurses help to ensure the patient's comfort as soon as possible by providing multidisciplinary cooperation in the management of complications that develop during this process. For this purpose, nurses need to carry out the necessary practices and precautions against the risk of developing PUR, which is one of the postoperative complications. In the recently published Nursing Regulation, the nurses' authority to manage PUR is clearly stated as "interventions to be implemented by a nursing decision" as "A nurse can decide independently or jointly with a physician to insert and remove a urinary catheter if she cannot eliminate urinary retention with the interventions she can apply", "Hot-cold application" intervention definition is clearly stated. Therefore, nurses evaluate the patient by reviewing the existing risk factors of the patient and surgical process during the perioperative period, providing emotional support for surgical stress, questioning perioperative fluid intake, informing the patient about the consumption of caffeine-containing drinks and plenty of water, monitor urine postoperatively, prefer non-invasive methods (listening to water sound, relaxation, bladder massage, mobilization, hot-cold application, ko mot/duck/sliders) primarily in case of PURE development, and invasive methods as a last resort (urinary catheterization, ensuring the necessary cooperation with the physician for interventional applications is one of the important responsibilities in process management. In the literature, it is stated that hot-cold application with bladder catheterization, one of the invasive methods, and hot-water insertion of the hand, massage, mobilization, promotion of liquid and coffee consumption, pelvic muscle exercise, and acupuncture are used in the management of PUR. In the studies conducted, the first postoperative urine output time was reduced by sacral massage in the management of PUR nurses; there was a rapid and permanent decrease in the development of PUR accompanied by the urination algorithm from 21% to 3% observed. However, 59.5% of patients with a hot compress applied to the bladder and 71.4% with cold application had urinary retention regressed; a significant difference in the severity of urinary retention was revealed by hot application; it is reported that urinary catheterization after the hot application is applied to only 3.9% of the patients. Based on these results, it is seen that the practices used by nurses to prevent and manage PUR have resulted in positive outcomes; the hot and cold practice has also made significant contributions to PUR management. For this purpose, it is envisaged that our study will contribute to the effective management of hot-cold application of PUR to the bladder in orthopedic surgery patients, to the minimum preference of invasive applications, to increasing the awareness of nurses about PUR management, and to the literature.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age,
* no urinary catheter inserted during the perioperative process, conscious and orientated,
* no renal disease (chronic kidney failure, nephropathy, kidney transplantation, prostate, urinary tract infection, history of stones in the urinary system)
* voluntary acceptance to participate in the study.

Exclusion Criteria:

* <18 years of age,
* intellectual disability or perception problem,
* communication disability,
* renal disease (chronic kidney failure, nephropathy, kidney transplantation, prostate, urinary tract infection, history of stones in the urinary system)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
physiological parameter, questionnaire | the first 6 hours of the postoperative period
  prevention of postoperative urinary retention by applying hot and cold to the bladder

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Yazici, Study Director — Assoc. Dr.
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asahara H, Inui M, Lotz MK. Tendons and Ligaments: Connecting Developmental Biology to Musculoskeletal Disease Pathogenesis. J Bone Miner Res. 2017 Sep;32(9):1773-1782. doi: 10.1002/jbmr.3199. Epub 2017 Jul 13. PMID 28621492
- [Background] Lum ZC, Pereira GC, Giordani M, Meehan JP. Top 100 most cited articles in orthopaedic surgery: An update. J Orthop. 2019 Dec 2;19:132-137. doi: 10.1016/j.jor.2019.11.039. eCollection 2020 May-Jun. PMID 32025120
- [Background] Casari FA, Navab N, Hruby LA, Kriechling P, Nakamura R, Tori R, de Lourdes Dos Santos Nunes F, Queiroz MC, Furnstahl P, Farshad M. Augmented Reality in Orthopedic Surgery Is Emerging from Proof of Concept Towards Clinical Studies: a Literature Review Explaining the Technology and Current State of the Art. Curr Rev Musculoskelet Med. 2021 Apr;14(2):192-203. doi: 10.1007/s12178-021-09699-3. Epub 2021 Feb 5. PMID 33544367
- [Background] Parry SM, Puthucheary ZA. The impact of extended bed rest on the musculoskeletal system in the critical care environment. Extrem Physiol Med. 2015 Oct 9;4:16. doi: 10.1186/s13728-015-0036-7. eCollection 2015. PMID 26457181
- [Background] LeBoff MS, Greenspan SL, Insogna KL, Lewiecki EM, Saag KG, Singer AJ, Siris ES. The clinician's guide to prevention and treatment of osteoporosis. Osteoporos Int. 2022 Oct;33(10):2049-2102. doi: 10.1007/s00198-021-05900-y. Epub 2022 Apr 28. PMID 35478046
- [Background] Waljee J, Zhong L, Baser O, Yuce H, Fox DA, Chung KC. The incidence of upper and lower extremity surgery for rheumatoid arthritis among Medicare beneficiaries. J Bone Joint Surg Am. 2015 Mar 4;97(5):403-10. doi: 10.2106/JBJS.N.00802. PMID 25740031
- [Background] Franke A, Bieler D, Wilms A, Hentsch S, Johann M, Kollig E. [Treatment of gunshot fractures of the lower extremity: Part 2: Procedures for secondary reconstruction and treatment results]. Unfallchirurg. 2014 Nov;117(11):985-94. doi: 10.1007/s00113-014-2636-x. German. PMID 25398508
- [Background] Moosavi Tekye SM, Alipour M. Comparison of the effects and complications of unilateral spinal anesthesia versus standard spinal anesthesia in lower-limb orthopedic surgery. Braz J Anesthesiol. 2014 May-Jun;64(3):173-6. doi: 10.1016/j.bjane.2013.06.014. Epub 2013 Oct 25. PMID 24907876
- [Background] Fernandez MA, Karthikeyan S, Wyse M, Foguet P. The incidence of postoperative urinary retention in patients undergoing elective hip and knee arthroplasty. Ann R Coll Surg Engl. 2014 Sep;96(6):462-5. doi: 10.1308/003588414X13946184902523. PMID 25198980
- [Background] David M, Arthur E, Dhuck R, Hemmings E, Dunlop D. High rates of postoperative urinary retention following primary total hip replacement performed under combined general and spinal anaesthesia with intrathecal opiate. J Orthop. 2015 Nov 18;12(Suppl 2):S157-60. doi: 10.1016/j.jor.2015.10.020. eCollection 2015 Dec. PMID 27047216
- [Background] Scholten R, Kremers K, van de Groes SAW, Somford DM, Koeter S. Incidence and Risk Factors of Postoperative Urinary Retention and Bladder Catheterization in Patients Undergoing Fast-Track Total Joint Arthroplasty: A Prospective Observational Study on 371 Patients. J Arthroplasty. 2018 May;33(5):1546-1551. doi: 10.1016/j.arth.2017.12.001. Epub 2017 Dec 13. PMID 29306574
- [Background] Kort NP, Bemelmans Y, Vos R, Schotanus MGM. Low incidence of postoperative urinary retention with the use of a nurse-led bladder scan protocol after hip and knee arthroplasty: a retrospective cohort study. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):283-289. doi: 10.1007/s00590-017-2042-5. Epub 2017 Sep 12. PMID 28900757
- [Background] Abdul-Muhsin HM, Jakob N, Cha S, Zhang N, Schwartz A, Navaratnam A, Khan A, Humphreys M. Incidence, Outcomes, and Prediction of Postoperative Urinary Retention After a Nonurologic Procedure. J Am Acad Orthop Surg Glob Res Rev. 2020 May;4(5):e1900149. doi: 10.5435/JAAOSGlobal-D-19-00149. PMID 33970584
- [Background] Balderi T, Mistraletti G, D'Angelo E, Carli F. Incidence of postoperative urinary retention (POUR) after joint arthroplasty and management using ultrasound-guided bladder catheterization. Minerva Anestesiol. 2011 Nov;77(11):1050-7. Epub 2011 May 11. PMID 21597444
- [Background] Bjerregaard LS, Bogo S, Raaschou S, Troldborg C, Hornum U, Poulsen AM, Bagi P, Kehlet H. Incidence of and risk factors for postoperative urinary retention in fast-track hip and knee arthroplasty. Acta Orthop. 2015 Apr;86(2):183-8. doi: 10.3109/17453674.2014.972262. Epub 2014 Oct 10. PMID 25301436
- [Background] Lior Y, Haim S, Katz I, Danino B, Bar-Yosef Y, Ekstein M. Postoperative Urinary Catheterization in Children Treated with or without Epidural Analgesia after Orthopedic Surgery: A Retrospective Review of Practice. Children (Basel). 2022 Aug 29;9(9):1316. doi: 10.3390/children9091316. PMID 36138625
- [Background] Zelmanovich A, Fromer DL. (2018). Urinary Retention after Orthopedic Surgery: Identification of Risk Factors and Management. J Clin Exp Orthop, 4(1):54. doi:10.4172/2471-8416.100054.
- [Background] Jackson J, Davies P, Leggett N, Nugawela MD, Scott LJ, Leach V, Richards A, Blacker A, Abrams P, Sharma J, Donovan J, Whiting P. Systematic review of interventions for the prevention and treatment of postoperative urinary retention. BJS Open. 2018 Nov 19;3(1):11-23. doi: 10.1002/bjs5.50114. eCollection 2019 Feb. PMID 30734011
- [Background] Cakmak M, Yildiz M, Akarken I, Karaman Y, Cakmak O. (2020). Risk Factors for Postoperative Urinary Retention in Surgical Population: A Prospective Cohort Study. J Urol Surg, 7(2): 144-148. doi: 10.4274/jus.galenos.2020.3544.
- [Background] Pomajzl AJ, Siref LE. (2022). Post-op Urinary Retention. https://www.ncbi.nlm.nih.gov/books/NBK549844/. 25 Kasım 2022.
- [Background] Agrawal K, Majhi S, Garg R. (2019). Post-operative urinary retention: Review of the literature. World J Anesthesiol, 8(1): 1-12. https://dx.doi.org/10.5313/wja.v8.i1.1.
- [Background] Irish Surgical Research Collaborative; Croghan SM, Fleming CA, Mohan HM, Harji D, Bolger JC, Elliott JA, Boland M, Lonergan PE, Dillon P, Quinlan DM, Winter DC. RETention of urine After INguinal hernia Elective Repair (RETAINER study I and II). Int J Surg Protoc. 2021 Apr 23;25(1):42-54. doi: 10.29337/ijsp.137. PMID 34013144
- [Background] Zheng C, Guo C. Intraoperative Urine Output Is Associated with Postoperative Outcome in Pediatric Population Undergone Major Abdominal Operations. Ther Clin Risk Manag. 2019 Dec 18;15:1453-1460. doi: 10.2147/TCRM.S228528. eCollection 2019. PMID 31908465
- [Background] Ceratti RDN, Beghetto MG. Incidence of urinary retention and relations between patient's complaint, physical examination, and bladder ultrasound. Rev Gaucha Enferm. 2021 Mar 12;42:e20200014. doi: 10.1590/1983-1447.2021.20200014. eCollection 2021. English, Portuguese. PMID 33886922
- [Background] World Health Organization (WHO), Improving the Quality of Health Services: Tools and Resources, 2018. Available from: https://apps.who.int/iris/bitstream/handle/10665/310944/9789241515085-eng.pdf. 14 Aralık 2022.
- [Background] Akhtar A, Macfarlane RJ, Waseem M. Pre-operative assessment and post-operative care in elective shoulder surgery. Open Orthop J. 2013 Sep 6;7:316-22. doi: 10.2174/1874325001307010316. eCollection 2013. PMID 24093051
- [Background] Official Gazette, Nursing Regulation, 2011. Number: 27910. https://www.resmigazete.gov.tr/eskiler/2011/04/20110419-5.html . December 14, 2022
- [Background] Malley A, Kenner C, Kim T, Blakeney B. The role of the nurse and the preoperative assessment in patient transitions. AORN J. 2015 Aug;102(2):181.e1-9. doi: 10.1016/j.aorn.2015.06.004. PMID 26227526
- [Background] McGarry JR, Pope C, Green SM. Perioperative nursing: maintaining momentum and staying safe. J Res Nurs. 2018 Dec;23(8):727-739. doi: 10.1177/1744987118808835. Epub 2018 Dec 7. PMID 34394495
- [Background] Urpo M, Eskola S, Suominen T, Roos M. (2021). Teamwork: a perspective of perioperative nurses. Central European Journal of Nursing and Midwifery, 12;430-440. doi:10.15452/cejnm.2021.12.0018.
- [Background] Yaban Simsek Z, Karaoz S. (2017). Effect of Nursing Interventions on Prevention and Management of Postoperative Urinary Retention for Patients with Orthopedic Surgery under Spinal Anaesthesia. International Journal of Caring Sciences, 10(1): 522-31.
- [Background] Wu AK, Auerbach AD, Aaronson DS. National incidence and outcomes of postoperative urinary retention in the Surgical Care Improvement Project. Am J Surg. 2012 Aug;204(2):167-71. doi: 10.1016/j.amjsurg.2011.11.012. Epub 2012 May 3. PMID 22560203
- [Background] Meska MH, Mazzo A, Jorge BM, Souza-Junior VD, Negri EC, Chayamiti EM. Urinary retention: implications of low-fidelity simulation training on the self-confidence of nurses. Rev Esc Enferm USP. 2016 Sep-Oct;50(5):831-837. doi: 10.1590/S0080-623420160000600017. English, Portuguese. PMID 27982403
- [Background] Uslu Y, Yavuz M. (2016). Urinary retention and management after surgery. New Journal of Urology, 11 (1): 48-53.
- [Background] Afazel MR, Jalali E, Sadat Z, Mahmoodi H. Comparing the effects of hot pack and lukewarm-water-soaked gauze on postoperative urinary retention; a randomized controlled clinical trial. Nurs Midwifery Stud. 2014 Dec;3(4):e24606. doi: 10.17795/nmsjournal24606. Epub 2014 Dec 29. PMID 25741518
- [Background] Dal U, Korucu AE, Eroglu K, Karatas B, Yalcin A. Sacral region massage as an alternative to the urinary catheter used to prevent urinary retention after cesarean delivery. Balkan Med J. 2013 Mar;30(1):58-63. doi: 10.5152/balkanmedj.2012.083. Epub 2013 Mar 1. PMID 25207070
- [Background] Leach D, Spaulding J, Thomas J, Conn C, Kutash M. The effect of caffeine on postoperative urinary retention after joint replacement surgery. Orthop Nurs. 2013 Sep-Oct;32(5):282-5. doi: 10.1097/NOR.0b013e3182a30184. PMID 24022423
- [Background] Zong J, You M, Li C. Effect of Kegel Pelvic Floor Muscle Exercise Combined with Clean Intermittent Self-catheterization on urinary retention after radical hysterectomy for cervical cancer. Pak J Med Sci. 2022 Mar-Apr;38(3Part-I):462-468. doi: 10.12669/pjms.38.3.4495. PMID 35480547
- [Background] Chen S, Sun H, Xu H, Zhang Y, Wang H. Effects of Acupuncture on Hospitalized Patients with Urinary Retention. Evid Based Complement Alternat Med. 2020 Jan 19;2020:2520483. doi: 10.1155/2020/2520483. eCollection 2020. PMID 32051686
- [Background] Brouwer TA, van Roon EN, Rosier PFWM, Kalkman CJ, Veeger N. Postoperative urinary retention: risk factors, bladder filling rate and time to catheterization: an observational study as part of a randomized controlled trial. Perioper Med (Lond). 2021 Jan 4;10(1):2. doi: 10.1186/s13741-020-00167-z. PMID 33397468
- [Background] Eldh AC, Joelsson-Alm E, Wretenberg P, Halleberg-Nyman M. Onset PrevenTIon of urinary retention in Orthopaedic Nursing and rehabilitation, OPTION-a study protocol for a randomised trial by a multi-professional facilitator team and their first-line managers' implementation strategy. Implement Sci. 2021 Jun 26;16(1):65. doi: 10.1186/s13012-021-01135-x. PMID 34174917
- [Background] Pierson M, Cretella B, Roussel M, Byrne P, Parkosewich J. A Nurse-Led Voiding Algorithm for Managing Urinary Retention After General Thoracic Surgery. Crit Care Nurse. 2022 Feb 1;42(1):23-31. doi: 10.4037/ccn2022727. PMID 35100628
- [Background] Seyedalangi H, Sajadi S A, Farsi Z, Mohamad Nejad E. (2015). The effect of warm compresses on urinary retention in male patients after cardiac catheterization hospitalized in military hospitals. MCS, 2(3):143-149. http://mcs.ajaums.ac.ir/article-1-86-en.html.
- [Background] Roudbari F. (2017). The effects of cold and hot compresses in the supra-pubic area on urinary retention in elderly patients after surgery. https://en.irct.ir/trial/19269. 13 Aralık 2022.
- [Background] COHEN J. The statistical power of abnormal-social psychological research: a review. J Abnorm Soc Psychol. 1962 Sep;65:145-53. doi: 10.1037/h0045186. No abstract available. PMID 13880271
- [Background] Meng MV, Tanagho EA. (2013). Physical Examination of the Genitourinary Tract. In: Smith and Tanagho's General Urology. McAninch JW, Lue TF. eds. Chapter 4. McGraw Hill.https://accessmedicine.mhmedical.com/content.aspx?bookid=508&sectionid=4108808. 16 December 2022.
- [Background] Nurcan C, Karadag M. (2015). Superficial Heat and Cold Applications in the Treatment of Knee Osteoarthritis. In: Osteoarthritis-Progress in Basic Research and Treatment. IntechOpen. https://doi.org/10.5772/60534.
- [Result] Gunay AE, Karaman I, Yazici A, Oner M, Ekici M, Kafadar I, et al. (2022). Distribution of Orthopedic Surgery Interventions: Evaluation of 6236 Cases. Erciyes Med J, 44(2): 173-7. doi:10.14744/etd.2021.05873.